CLINICAL TRIAL: NCT00262691
Title: Investigation of Genetic Risk of Cardiovascular Disease in Prospective Cohort Study, the Kitanagoya Genome (KING) Study for the Local Residents of Kitanagoya, Japan
Brief Title: Investigation of Genetic Risk of Cardiovascular Disease in Prospective Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nagoya University (Other)
Collaborators: Aichi Gakuin University (Other)
Other Study IDs: NU-05-G-0001
Record Dates: First submitted 2005-12-06; First posted 2005-12-07 (Estimated); Last update posted 2007-09-21 (Estimated); Status verified 2007-09

CONDITIONS: Healthy; Coronary Disease; Myocardial Infarction; Cerebral Infarction
MeSH Terms: conditions — Coronary Disease; Myocardial Infarction; Cerebral Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Cardiovascular disease is a complex multifactorial and polygenic disorder that is thought to result from an interaction between a person's genetic make up and various environmental factors. Although many studies have revealed that several genetic variants increase the risk of cardiovascular disease, the results of these studies remain controversial. The purpose of this study is to identify polymorphisms that confer susceptibility to cardiovascular disease and to clarify the adequacy of reported susceptibility gene polymorphisms. To complete this purpose, we will prospectively study over 5,000 local residents in whom relationship between these polymorphisms and occurrence of cardiovascular disease over 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects who undergo community-based annual health check in Kitanagoya city

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7000 (Estimated)
Dates: Start 2005-05

CONTACTS AND LOCATIONS:
Overall Officials: Mitsuhiro Yokota, MD, PhD, Study Chair — Department of Genome Science, School o Dentistry, Aichi-Gakuin University
Locations (1):
- Department of Genome Science, School of Dentistry, Aichi-Gakuin University, Nagoya, Aichi-ken, Japan

REFERENCES:
- [Derived] Ohashi Y, Ichihara S, Yamamoto K, Kitamura Y, Matsubara T, Beppo R, Kinoshita F, Kato TS, Toyoda Y, Kawamura Y, Matsuo H, Ichida K, Yokota M, Nakatochi M. Proteomic footprint of serum urate concentration and urate transporter ABCG2 dysfunctional polymorphism: a cross-sectional study. RMD Open. 2026 Jan 27;12(1):e006414. doi: 10.1136/rmdopen-2025-006414. PMID 41592914
- [Derived] Nakatochi M, Ichihara S, Yamamoto K, Naruse K, Yokota S, Asano H, Matsubara T, Yokota M. Epigenome-wide association of myocardial infarction with DNA methylation sites at loci related to cardiovascular disease. Clin Epigenetics. 2017 May 15;9:54. doi: 10.1186/s13148-017-0353-3. eCollection 2017. PMID 28515798
- [Derived] Nakatochi M, Miyata S, Tanimura D, Izawa H, Asano H, Murase Y, Kato R, Ichihara S, Naruse K, Matsubara T, Honda H, Yokota M. The ratio of adiponectin to homeostasis model assessment of insulin resistance is a powerful index of each component of metabolic syndrome in an aged Japanese population: results from the KING Study. Diabetes Res Clin Pract. 2011 Jun;92(3):e61-5. doi: 10.1016/j.diabres.2011.02.029. Epub 2011 Mar 31. PMID 21458098
- [Derived] Tanimura D, Shibata R, Izawa H, Hirashiki A, Asano H, Murase Y, Miyata S, Nakatochi M, Ouchi N, Ichihara S, Yasui K, Yoshida T, Naruse K, Matsubara T, Yokota M. Relation of a common variant of the adiponectin gene to serum adiponectin concentration and metabolic traits in an aged Japanese population. Eur J Hum Genet. 2011 Mar;19(3):262-9. doi: 10.1038/ejhg.2010.201. Epub 2010 Dec 8. PMID 21150884
- [Derived] Asano H, Izawa H, Nagata K, Nakatochi M, Kobayashi M, Hirashiki A, Shintani S, Nishizawa T, Tanimura D, Naruse K, Matsubara T, Murohara T, Yokota M. Plasma resistin concentration determined by common variants in the resistin gene and associated with metabolic traits in an aged Japanese population. Diabetologia. 2010 Feb;53(2):234-46. doi: 10.1007/s00125-009-1517-2. Epub 2009 Sep 1. PMID 19727657